CLINICAL TRIAL: NCT05279872
Title: A Study of Zanubrutinib in Patients With Primary Immune Thrombocytopenia (ITP)
Brief Title: A Study of Zanubrutinib in Patients With ITP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking University Institute of Hematology, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKU-ITP032
Record Dates: First submitted 2022-01-24; First posted 2022-03-15 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Immune Thrombocytopenia; Bruton Tyrosine Kinase
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinib (Experimental): Zanubrutinib 80mg po qd 6 weeks
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib 80mg po qd 6 weeks

SUMMARY:
This project was undertaken to evaluate the efficacy and safety of BTK inhibitor Zanubrutinib for the secondary treatment of adults with primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators are undertaking a prospective trial of 10 adults with ITP in China. Zanubrutinib is administered as 80 mg po. qd for 6 weeks. Platelet count, bleeding and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary refractory ITP
* Platelet counts <30×10^9/L or with bleeding symptoms
* Willing and able to sign written informed consent

Exclusion Criteria:

* Secondary thrombocytopenia
* Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 6 months before the screening visit
* HIV infection or hepatitis B virus or hepatitis C virus infections
* Malignancy
* Severe medical condition (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
* Nursing or pregnant patients
* Patients who are deemed unsuitable for the study by the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Overall response (OR) | 6 weeks
  The maintenance of platelet count ≥ 30 x 10^9/L, at least 2-fold increase of the baseline count, the absence of bleeding, and no need for rescue medication at the 6-week follow-up.

SECONDARY OUTCOMES:
Complete response (CR) | 6 weeks
  Complete response (CR) was defined as platelet count more than 100,000 per cubic millimeter and absence of bleeding.
Time to response | 6 weeks
  The time from starting treatment to time of achievement of Response.
Bleeding events | 6 weeks
  The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Side Effects | 6 weeks
  Potential side effects include leukopenia, nausea and diarrhea, infectious diseases, etc .

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University People's Hospital, Peking University Institute of Hematology, National Clinical Research Center for Hematologic Disease, Beijing Key Laboratory of Hematopoietic Stem Cell Transplantation, Collaborative Innovation Center of Hematology
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang QS, Fu HX, Wang CC, Zhu XL, He Y, Wu J, Chen Q, Zhao P, An ZY, Liu KY, Huang XJ, Zhang XH. Efficacy and Safety of the Bruton's Tyrosine Kinase Inhibitor Zanubrutinib in Immune Thrombocytopenia. Am J Hematol. 2025 Aug;100(8):1314-1322. doi: 10.1002/ajh.27718. Epub 2025 May 20. PMID 40391880